CLINICAL TRIAL: NCT05421247
Title: A Descriptive Study on Children With COVID-19 Admitted at Isolation Unit of Assiut University Children Hospital
Brief Title: A Study on Children With COVID-19 Admitted at Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abd Elaal Ahmed, resident at Assiut University Children Hospital, Assiut University
Other Study IDs: COVID-19 in children
Record Dates: First submitted 2022-06-15; First posted 2022-06-16 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: children; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of study is to: 1-describe demographic and clinical data of children infected with COVID-19 admitted at isolation unit of Assiut university children hospital 2- assess the risk factors responsible for complications of COVID-19 in children 3-assess the outcome of COVID-19 in children admitted at AUCH.

DETAILED DESCRIPTION:
In December 2019, reports emerged of a cluster of cases of pneumonia of unknown cause in Wuhan, China, culminating in the identification of a novel coronavirus on 12 January 2020, denoted as severe acute respiratory syndrome coronavirus 2 (SARSCoV-2), and the associated disease as coronavirus disease 2019 (COVID-19) (1).

Some cases of infection in children have also been reported (2) the symptoms of pediatric COVID-19 are mild, the decrease in lymphocytes is not obvious and severe cases are rare. Initially, children comprised between 1% and 2% of the laboratory-confirmed SARSCoV-2 detections among people in China (3), Italy (4), and the United States (5). Initial reports from (CDC) noted the following age distributions: 15-17 years (32%), 10-14 years (27%), 5-9 years (15%), 1-4 years (11%), and <1 year (15%), with a median age of 11 years (5).

Diagnosis of COVID-19 will depend on the clinical presentation of the case and on laboratory test as well as radiological finding. The cases will be stratified according to these collective data to different grades of severity (6). Investigations for suspected case: CBC and radiology, to confirm diagnosis: Nasopharyngeal swab for PCR and to assess severity: Serum ferritin, D dimer, LDH, and CRP. (7) Current treatment for COVID-19 is mainly supportive care (8).The decision of the site of management either at home or in hospital depends on the clinical presentation, requirement for supportive care, potential risk factors for severe disease, and the ability of the patient to self-isolate at home(9) (10).

ELIGIBILITY:
Inclusion Criteria:

* All children (up to 18 years) diagnosed with COVID-19 admitted at Isolaton Unit of Assiut university children hospital through the period from 1st January 2021 to 31st December 2022

Exclusion Criteria:

* Clinically suspected patients approved by CT chest and PCR not infected with COVID-19.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children (up to 18 years) diagnosed with COVID-19 admitted at Isolaton Unit of Assiut university children hospital through the period from 1st January 2021 to 31st December 2022
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
to describe demographic and clinical data of children infected with COVID-19 admitted at isolation unit of Assiut university children hospital | Baseline
  to describe demographic data (age ,sex ,residence , socioeconomics,...etc.) and length of hospital stay

SECONDARY OUTCOMES:
to assess the risk factors responsible for complications of COVID-19 in children. | Baseline
  History of contact with patients positive for COVID-19, If associated comorbidities for example DM, immune deficiency and chronic kidney disease
to assess the outcome of COVID-19 in children admitted at AUCH | Baseline
  to assess the number of cases with complete recovery , the number of deaths and the cases with different complications as respiratory failure , renal failure ...etc and normalization of lab. data as(lymphocytic count , D- dimer , CRP ) and CORAD staging on chest CT

CONTACTS AND LOCATIONS:
Overall Officials: Nagla H. Ibrahim, professor, Study Director

REFERENCES:
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Dong Y, Mo X, Hu Y, Qi X, Jiang F, Jiang Z, Tong S. Epidemiology of COVID-19 Among Children in China. Pediatrics. 2020 Jun;145(6):e20200702. doi: 10.1542/peds.2020-0702. Epub 2020 Mar 16. PMID 32179660
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020 Apr 14;323(14):1335. doi: 10.1001/jama.2020.4344. No abstract available. PMID 32181795
- [Background] CDC COVID-19 Response Team. Coronavirus Disease 2019 in Children - United States, February 12-April 2, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 10;69(14):422-426. doi: 10.15585/mmwr.mm6914e4. PMID 32271728
- [Background] [6] Masoud H, Elassal G, Zaky S, Baki A, Ibrahim H, Amin W, et al. Management Protocol for COVID-19 Patients Version 1.4/30th May 2020 Ministry of health and population (MOHP), Egypt. 2020.
- [Background] [7] Mostafa A, Abdalbaky A, Fouda E, Shaaban H, Elnady H, Hassab-Allah M et al. Practical approach to COVID-19: an Egyptian pediatric consensus. Egyptian Pediatric Association Gazette. 2020;68(1).
- [Background] Klein JD, Koletzko B, El-Shabrawi MH, Hadjipanayis A, Thacker N, Bhutta Z. Promoting and supporting children's health and healthcare during COVID-19 - International Paediatric Association Position Statement. Arch Dis Child. 2020 Jul;105(7):620-624. doi: 10.1136/archdischild-2020-319370. Epub 2020 May 7. No abstract available. PMID 32381517
- [Background] Chen ZM, Fu JF, Shu Q, Chen YH, Hua CZ, Li FB, Lin R, Tang LF, Wang TL, Wang W, Wang YS, Xu WZ, Yang ZH, Ye S, Yuan TM, Zhang CM, Zhang YY. Diagnosis and treatment recommendations for pediatric respiratory infection caused by the 2019 novel coronavirus. World J Pediatr. 2020 Jun;16(3):240-246. doi: 10.1007/s12519-020-00345-5. Epub 2020 Feb 5. PMID 32026148